CLINICAL TRIAL: NCT03360344
Title: Effects on Occupational Performance Through Dorsal Application of Kinesio Tape for Musculoskeletal Disorder - Carpal Tunnel Syndrome
Brief Title: Non-surgical Intervention for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Heather Javaherian-Dysinger, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 5170437
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Carpal Tunnel Syndrome, Susceptibility to
Keywords: carpal tunnel syndrome, pain, numbness, kinesio tape
MeSH Terms: conditions — Carpal Tunnel Syndrome; Pain; Hypesthesia

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled trial
Who Masked: Participant
Masking Description: Participants do not know which group they will be randomly assigned
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Kinesio Tape (Experimental): Dorsal application of Kinesio Tape to the affected extremity: Approximately 12 inches of Kinesio tape will be applied from the musculotendinous junction of the participant's forearm over digits 1 and 5. Two - 2 inch strips of Kinesio Tape will be applied to the participant's wrists over the volar and dorsal aspects. The Kinesio Tape will remain in place for three days, with the participants returning for skin check by the researchers and re-application by the researchers four times during the course of the study.
  A tape removal form will be provided should the participants want to remove it prior to the next visit.
  Interventions: Device: Kinesio 12 inch Tape
- Control group (Sham Comparator): Approximately 4 inch strip of Kinesio Tape will be applied to the scapular spine of the same side as the affected extremity. The Kinesio Tape will remain in place for three days, with the participants returning for skin check by the researchers and re-application four times during the course of the study by the researcher. A tape removal form will be provided should the participants want to remove it prior to the next visit.
  Interventions: Device: Kinesio 4 inch Tape
- Standard of Care (Active Comparator): Currently, the standard of care is a general cock-up splint and lumbrical exercises. A general cock-up splint will be supplied, fitted, and checked on each of the four return visits by the researchers. Lumbrical exercises are also used and consist of active joint ranges for the wrist and hand. The exercises will be demonstrated by the researchers for 3-sets of 10 times each, daily, to be recorded in a log by the participants.
  Interventions: Device: Cock up Splint and Lumbrical exercises

INTERVENTIONS:
Device: Kinesio 12 inch Tape — Kinesio Tape approximately 12-inch strip will be applied to the dorsal surface of the forearm of the affected side for three-day increments over three weeks of the study.
  Arms: Kinesio Tape
Device: Kinesio 4 inch Tape — Kinesio Tape for the control group will be a 4 inch Kinesio Tape applied to the scapular spine for three day increments over three weeks of the study.
  Arms: Control group
Device: Cock up Splint and Lumbrical exercises — A general cock-up splint will be supplied, fitted, and checked on each of the four return visits by the researchers. Lumbrical exercises are also used and consist of active joint ranges for the wrist and hand. The exercises will be demonstrated by the researchers for 3-sets of 10 times each, daily, to be recorded in a log by the participants.
  Arms: Standard of Care

SUMMARY:
This randomized controlled trial graduate student research study will explore the effect of non-surgical intervention of the dorsal application of Kinesio Tape for carpal tunnel syndrome, and forearm wrist hand pain.

DETAILED DESCRIPTION:
This randomized controlled trial graduate student research study will explore the effect of non-surgical intervention of the dorsal application of Kinesio Tape for carpal tunnel syndrome, and forearm wrist hand pain. Little evidence exists for an effective non-surgical intervention. Semi-structured interviews will be conducted to explore changes in occupational performance and compliance in order to understand if Kinesio Tape contributed to results and if so, how the participants perceived the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years of age
* Fluent in English
* Report signs and symptoms of carpal tunnel syndrome
* Pain, numbness, and tingling of the forearm, wrist, or hand, which worsen at night
* Demonstrate positive Phalen's Test or Tinel's Test of the affected extremity

Exclusion Criteria:

* Currently receiving treatment for carpal tunnel syndrome
* History of surgical carpal tunnel release
* Pregnant
* Diabetes not controlled by medication
* Radiculopathy ie: cervical radiculopathy, diabetic radiculopathy
* Thoracic outlet syndrome
* Allergy to adhesives or compromised skin integrity
* Past history of traumatic event, surgery, or congenital impairment of the forearm, wrist, or hand

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grenith Zimmerman, PhD, Study Chair — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-four (44) participants and sixty-eight (68) wrists were enrolled in the study. Some participants had bilateral involvement whereas other participants only had one wrist that was involved.
Units Other Than Participants: wrist
Groups:
- Kinesio Tape: Dorsal application of Kinesio Tape to the affected extremity: Approximately 12 inches of Kinesio tape will be applied from the musculotendinous junction of the participant's forearm over digits 1 and 5. Two - 2 inch strips of Kinesio Tape will be applied to the participant's wrists over the volar and dorsal aspects. The Kinesio Tape will remain in place for three days, with the participants returning for skin check by the researchers and re-application by the researchers four times during the course of the study.
  A tape removal form will be provided should the participants want to remove it prior to the next visit.
  Kinesio 12 inch Tape: Kinesio Tape approximately 12-inch strip will be applied to the dorsal surface of the forearm of the affected side for three-day increments over three weeks of the study.
Period: Overall Study
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Started (Analysis was completed on 68 wrists (units of study)) | 15; 25 wrist | 16; 20 wrist | 13; 23 wrist
Completed (Analysis was completed on 68 wrists (units of study)) | 15; 25 wrist | 15; 19 wrist | 12; 22 wrist
Not Completed | 0; 0 wrist | 1; 1 wrist | 1; 1 wrist
Not completed — Withdrawal by Subject | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline randomized participants (n = 44) and baseline wrists as the unit of measure was (n = 68). A percentage of participants had bi-lateral symptomatic wrists.
  Analyzed randomized participants (n = 42) and analyzed wrists (n = 66). Two (2) participants voluntarily withdrew.
Units Other Than Participants: wrists
Groups:
- Total: Total of all reporting groups
Arm/Group | Kinesio Tape | Standard of Care | Control Group | Total
Number analyzed (Participants) | 15 | 15 | 12 | 42
Number analyzed (wrists) | 25 | 19 | 22 | 66
Age, Continuous [Median (Full Range); unit: years] — Population: Baseline randomized participants (n = 44) and baseline wrists as the unit of measure was (n = 68). A percentage of participants had bi-lateral symptomatic wrists.
  Analyzed randomized participants (n = 42) and analyzed wrists (n = 66). Two (2) participants voluntarily withdrew
  years | 28 [23 to 67] | 28 [21 to 57] | 45 [23 to 76] | 29.5 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline randomized participants (n = 44) with baseline wrists as the unit of measure represented was (n = 68).
  Analyzed randomized participants (n = 42) and analyzed wrists as units of measure were (n = 66).
  Participants
    Female | 13 | 14 | 11 | 38
    Male | 2 | 1 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Please note that 2 subjects voluntarily withdrew from the study therefore the demographic table is based on n=42. Population: Randomized participants at baseline (n = 44) with wrists as the unit of measure was (n = 68).
  Analyzed participants was (n = 42) and analyzed wrists (n = 66)
  Participants
    African American | 0 | 0 | 1 | 1
    Asian | 4 | 3 | 2 | 9
    Caucasian or White | 7 | 8 | 7 | 22
    Latino/Hispanic | 4 | 2 | 1 | 7
    Non-Hispanic | 0 | 0 | 1 | 1
    Mixed | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants] — Population: Two participants voluntarily withdrew from the study, One from the "Standard Care" group and one from the "Control Group"
  participants
    United States | 15 | 15 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Rating Scale (NRS Pain)
Description: Numerical Pain Rating Scale (NRS Pain) involves patient circling a number from 0-10 with "0" meaning no pain and "5" moderate pain, and "10" is worst possible pain. The NRS is a segmented numeric scale, which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain. Higher scores indicate greater pain intensity.
Time Frame: change between baseline and 3 weeks
Measure: Median (Full Range); unit: score on a scale
Units Other Than Participants: Wrists
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Number analyzed (Participants) | 15 | 15 | 12
Number analyzed (Wrists) | 25 | 19 | 22
score on a scale
  Forearm | 0.01 [0 to 7] | .17 [0 to 7] | .30 [0 to 7]
  Wrist | .005 [0 to 8] | .11 [0 to 8] | .43 [0 to 9]
Statistical Analysis 1: Comparison: Kinesio Tape vs Standard of Care vs Control Group; statistical analysis for wrist; Test type: Other — non-parametric tests were used as data was not normally distributed; p = 0.48, Wilcoxan signed Rank
Statistical Analysis 2: Comparison: Kinesio Tape vs Standard of Care vs Control Group; statistical analysis for forearm; Test type: Other — nonparametric test were used as the distribution was not normal; p = .99, Wilcoxan Signed Rank

2. Primary Outcome: Visual Analog Scale for Pain (VAS Pain)
Description: The Visual Analogue Scale (VAS) is unidimensional measure of pain intensity, which has been widely used in diverse adult populations. The VAS measures participants perception of pain on a continuous scale. Individuals place a mark on a 10cm-long line. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. These are measured every 3 days for 3 weeks from baseline in the forearm, wrist and fingers.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Wrists
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Number analyzed (Participants) | 15 | 15 | 12
Number analyzed (Wrists) | 25 | 19 | 22
score on a scale
  Forearm | 18.64 (3.88) | 12.8 (4.12) | 15.2 (4.45)
  Wrist | 21.4 (4.65) | 32.6 (4.96) | 24.2 (5.3)
Statistical Analysis 1: Comparison: Kinesio Tape vs Standard of Care vs Control Group; statistical analysis for forearm; Test type: Other; p = .001, ANOVA
Statistical Analysis 2: Comparison: Kinesio Tape vs Standard of Care vs Control Group; statistical analysis for wrist; Test type: Other; p = .001, ANOVA

3. Secondary Outcome: Grip Strength and Pinch Strength
Description: Grip strength is measured by Jamar Dynamometer hydraulic gauge following standard protocol. A Jamar hydraulic pinch meter gauge is used to measure finger strength in the following positions: Lateral pinch, pad to pad, and 3 Jaw-chuck pinch positions are used. Grip and pinch strength will be measured every 3 days for 3 weeks from baseline.
Time Frame: change between baseline and 3 weeks
Measure: Mean (Standard Error); unit: lbs
Units Other Than Participants: wrists
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Number analyzed (Participants) | 15 | 15 | 12
Number analyzed (wrists) | 25 | 19 | 22
lbs
  Grip | 55.47 (3.7) | 64.8 (4.0) | 52.7 (4.3)
  pinch | 12.2 (.95) | 12.4 (.95) | 11.8 (1.1)
Statistical Analysis 1: Comparison: Kinesio Tape vs Standard of Care vs Control Group; Test type: Other; p = .06, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Boston Carpal Tunnel Questionnaire Symptom Severity (BCTQ SS)
Description: The Boston Carpal Tunnel Questionnaire (BCTQ SS) is a standardised, patient-based outcome measure of symptom severity in patients with carpal tunnel syndrome. The questionnaire has 11 questions and uses a five-point rating scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability. It is measured every 3 days for 3 weeks from baseline.
Time Frame: change between baseline and 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: wrists
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Number analyzed (Participants) | 15 | 15 | 12
Number analyzed (wrists) | 25 | 19 | 22
score on a scale | 1.9 (.04) | 2.0 (.04) | 2.0 (.04)
Statistical Analysis 1: Comparison: Kinesio Tape vs Standard of Care vs Control Group; Test type: Other; p = .01, ANCOVA

5. Secondary Outcome: Boston Carpal Tunnel Questionnaire Functional Scale (BCTQ FS)
Description: The Boston Carpal Tunnel Questionnaire Functional Scale (BCTQ FS) is self report 8-item questionnarie on functional activities for individuals with carpal tunnel, which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability. It is measured every 3 days for 3 weeks from baseline.
Time Frame: 3-weeks
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Wrists
Arm/Group | Kinesio Tape | Standard of Care | Control Group
Number analyzed (Participants) | 15 | 15 | 12
Number analyzed (Wrists) | 25 | 19 | 22
score on a scale | 1.5 (.12) | 1.8 (.13) | 1.7 (.14)
Statistical Analysis 1: Comparison: Kinesio Tape vs Standard of Care vs Control Group; Test type: Other; p = .001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 3-weeks
Arm/Group | Kinesio Tape | Control Group | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03360344/Prot_SAP_000.pdf